CLINICAL TRIAL: NCT00133029
Title: The Timing of Prophylactic Antibiotics in Cesarean Section and the Risk of Post-operative Febrile Morbidity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 705719
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Cesarean Section

INTERVENTIONS:
Drug: Timing of prophylactic antibiotic administration

SUMMARY:
The purpose of this study is to determine whether the timing of prophylactic antibiotic administration for cesarean section (immediate preoperative versus intraoperative administration) impacts the rate of postoperative febrile morbidity. The specific aim of the project is to test the hypothesis that preoperative antibiotic administration will decrease the rate of composite postoperative febrile morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 36 weeks
* Ability to understand requirements of the study
* Elective/non-emergent cesarean section selected as route of delivery by treating physicians

Exclusion Criteria:

* Known fetal anomaly
* Exposure to antibiotics within 7 days of admission, including intrapartum group B streptococcal (GBS) prophylaxis
* Emergent cesarean delivery (i.e. for fetal distress, maternal distress, obstetric hemorrhage)
* Overt maternal intrapartum infection requiring antibiotics
* Prolonged rupture of membranes (>18 hours)

Sex: Female
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A. Macones, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States